CLINICAL TRIAL: NCT06263335
Title: Impact of Mindfulness Based Therapeutic Intervention on Psychological Distress, Suicidal Ideation and Non-Suicidal Self Injury Among Young Adults: A Randomized Controlled Trial
Brief Title: MBI for Psychological Distress, SI and NSSI Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Sadia Sohail, Student, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fatima Jinnah Women University
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Psychological Distress; Suicidal Ideation; Non-Suicidal Self Injury
Keywords: Mindfulness Based Intervention; Psychological Distress; Suicidal Ideation; Non-Suicidal Self Injury
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Receiving Mindfulness Based Intervention) (Experimental): after the young adults have been randomized into interventional and control groups based on high levels of psychological distress, SI and NSSI, n=30 participants from this group would receive the mindfulness based intervention.
  Interventions: Other: Mindfulness Based Stress Reduction Intervention
- Control Group (No Intervention) (No Intervention): A wait list control group of n=30 randomized participants from the initial cohort would be in this group and receive no intervention, until the trial is completed.

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction Intervention — During an eight-week intervention period, clients were to engage in mindfulness practices lasting between 45 minutes to an hour each session. The intervention would incorporate various components of the Mindfulness-Based Stress Reduction (MBSR) program, including mindfulness of the present moment, body scans, mindful eating, walking meditation, yoga exercises, and discussions on applying mindfulness to everyday experiences and stress management. Sessions would typically range from 30 to 90 minutes per week, with an additional full-day retreat session towards the end of the program. In addition to mindfulness practice, participants were to receive teachings on stress management and its application to interpersonal and daily life situations.
  Arms: Interventional Group (Receiving Mindfulness Based Intervention)

SUMMARY:
Designed to measure the impact of Mindfulness Based Intervention on depression, anxiety, stress, psychological distress, Suicidal Ideation, Non-Suicidal Self Injury urge and Mindfulness in young adults. Those individuals who agree to participate in the trial and identified with high levels of psychological distress and Suicidal Ideation, randomly divided into interventional (n=30) and control (n=30) groups. The Mindfulness Based Stress Reduction intervention then administered to the interventional group for eight weeks and pre and post intervention assessment done for both the groups.

DETAILED DESCRIPTION:
Study assessment measures:

* Informed consent form
* Demographic questionnaire
* Screener questions form
* Assessment instruments:
* Depression Anxiety and Stress Scale (DASS-21)
* Suicide Ideation Scale (SIS)
* Alexian Brothers Urge to Self Injure Scale (ABUSI)
* Mindfulness Attention Awareness Scale

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-24, of any gender, who consented to participate and could comprehend English (the language of the questionnaires).
* Selected respondents from the initial survey were included based on specific criteria:
* Willingness to continue participation.
* Unmarried status.
* Pursuing education (Bachelors, Masters, or Ph.D.) , Pakistan.
* Non-hosteller and unemployed.
* Residing with both parents.
* Affirmative response to screener questions about suicidal ideation (SI) and non-suicidal self-injury (NSSI).
* High scores on psychological distress and SI scales.

Exclusion Criteria:

* Participants failing to meet inclusion criteria or falling under the following categories were excluded:
* Non-students.
* History of present or past psychiatric illness, with recent medication or treatment within the past year.
* Presence of debilitating physical diseases or disabilities. Involvement in or history of substance use.
* Long-term medication for any condition, as these factors could impact study results.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Psychological Distress | 8-12 weeks
  This refers to the overall level of emotional suffering or discomfort experienced by individuals, often encompassing symptoms of depression, anxiety, and stress. In this study, psychological distress serves as a primary outcome measure because it is a key variable being assessed in relation to the intervention's efficacy.
Suicidal Ideation | 8-12 weeks
  Suicidal ideation involves thoughts or ideas about engaging in behaviors intended to end one's life. As a primary outcome measure, assessing suicidal ideation is crucial in understanding the impact of the intervention on the participants' mental health and risk of self-harm.
Non-Suicidal Self-Injury (NSSI) | 8-12 weeks
  NSSI refers to deliberate, self-inflicted harm to one's body without suicidal intent, such as cutting or burning oneself. It is an essential primary outcome measure in this study because it directly relates to the intervention's effectiveness in reducing self-harming behaviors among participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Women University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Within the ethical considerations, results of research would be shared via research publications.
Supporting Information: CSR
Time Frame: When research is published.
Access Criteria: Through open access journal publications.